CLINICAL TRIAL: NCT06078917
Title: Endovascular Treatment for Acute Ischemic Stroke in Chinese Municipal and County Hospitals： A "Real World" Study-ETERNITY Registry
Brief Title: Endovascular Treatment for AIS in Chinese Municipal and County Hospitals： A "Real World" Study-ETERNITY Registry
Status: Completed | Type: Observational
Sponsor: Wen-huo Chen (Other)
Responsible Party: Sponsor-Investigator, Wen-huo Chen, Endovascular Treatment for Acute Ischemic Stroke in Chinese Municipal and County Hospitals： A "Real World" Study-ETERNITY Registry, Zhangzhou Municipal Hospital
Organization: Zhangzhou Municipal Hospital (Other)
Other Study IDs: A "Real world" study-ETERNITY
Record Dates: First submitted 2023-10-05; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Endovascular Treatment
Keywords: Endovascular Treatment; acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the Endovascular Treatment difference between Chinese city and country hospital.

DETAILED DESCRIPTION:
Endovascular Treatment for AIS in Chinese Municipal and County Hospitals： A "Real World" Study-ETERNITY Registry is an academic , independent, pragmatic , prospective , multicenter , observational registry study . Patients with acute ischemic stroke caused by anterior circulation intracranial large vessel occlusion and receiving EVT were included. Patients were divided into primary stroke center (county hospital) and senior stroke center (city hospital) groups. Acute ischemic stroke (AIS) workflow, EVT procedural details and clinical outcome were compared in two groups. The aim of the study was to explore the EVT difference in Chinese city and county hospital.

ELIGIBILITY:
Inclusion Criteria:

(1) age ≥18 years; (2) diagnosis of AIS caused by imaging-confirmed intracranial LVO, including isolated cervical internal carotid artery or tandem occlusion, intracranial internal carotid artery, middle cerebral artery (M1/M2), anterior cerebral artery (A1/A2); (3) initiation of any type of EVT, including mechanical thrombectomy, emergent angioplasty via balloon or/and stent; (4).Onset-to-presentation time with 24 hours; (5).Patients whose onset-to-presentation time surpass 6 hours should had CTP and fulfill with DAWN[6] or DEFUSE's[7] criteria.

Exclusion Criteria:

(1) Without follow up outcome; (2) posterior circulation stroke;(3)no evidence of LVO on angiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke caused by anterior circulation intracranial large vessel occlusion and receiving EVT were included.
Sampling Method: Probability Sample
Enrollment: 1196 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
The modified Rankin Scale score at 90 days | 90 days
  The range of the modified Rankin Scale is from 0 to 6. A higher score indicates a worse outcome.
  0-No symptoms; 1-No significant disability; 2-Slight disability; 3-Moderate disability; 4-Moderately severe disability; 5-Severe disability; 6-Dead.
Baseline CT/magnetic resonance and CT angiography/magnetic resonance angiography imaging, digital subtraction angiography | 90 days
  Radiological assessment included ASPECTS ，location of occlusion site, presence of underlying ICAS ，or exist microcatheter "First-Pass Effect".
Successful reperfusion | 90 days
  Successful reperfusion was defined as eTICI ≥2b

CONTACTS AND LOCATIONS:
Overall Officials: Wen-huo Chen, bachelor, Principal Investigator — Zhangzhou Affiliated Hospital to Fujian Medical University , Fujian ,China
Locations (1):
- Zhangzhou Municipal Hospital, Zhangzhou, Fujian, China